CLINICAL TRIAL: NCT04272723
Title: Management of Venous Thromboembolism in France: a National Survey Among Vascular Medicine Physicians
Acronym: Observ-MTEV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0014
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Survey; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Anticoagulant
Keywords: Survey; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Anticoagulant; Clinical Practice; Therapeutic management
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VMP members of the SFMV: VMP (vascular medicine physicians) members of the SFMV (French Society of Vascular Medicine )
- VMP registered as willing to do medical research: VMP (vascular medicine physicians) registered as willing to do medical research

SUMMARY:
In France, venous thromboembolic (VTE) disease is usually managed by vascular medicine physicians (VMP). The national OPTIMEV study, conducted more than 12 years ago among VMP practicing in hospital and in the community described the management of VTE in routine clinical practice. Since then a large number of practice changing studies have been published. This includes trials that have validated the use of direct oral anticoagulants (DOAC), the new standard of care of VTE, as per new national and international guidelines. Management of VTE in 2019 appears to be significantly different from the one that prevailed more than 10 years ago when the last national survey was conducted. It is therefore important to have an update on the routine clinical practice management of VTE by VMP. In this perspective the investigators aim to conduct a national survey among VMP practicing in France

ELIGIBILITY:
Inclusion Criteria:

* vascular medicine physicians who are active members of the SFMV (French Society of Vascular Medicine)
* vascular medicine physicians registered as willing to do medical research

Exclusion Criteria:

* vascular medicine physicians who refuse to provide consent
* vascular medicine physicians who are retired
* non-practicing vascular medicine physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular medicine physicians (VMP) practicing in the hospital and in the community settings.
  Participating VMP will prospectively collect data on the management of incident venous thromboembolic (VTE) disease cases.
  After that, vascular medicine physicians will answer a phone questionnaire on their general VTE management
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Inter-practician variability of clinical care of venous thromboembolic in routine clinical practice | up to 3 months after inclusion
  The variation in venous thromboembolic management in routine clinical practice is assessed by analysing the management of the 5 consecutive acute venous thromboembolic patients reported by each participating physician

SECONDARY OUTCOMES:
Inter-practician variability of clinical care of venous thromboembolic according to patient age | up to 6 months after inclusion
  patient characteristics are : cancer, extreme body weight, severe renal impairment, elderly or pregnant patients, high bleeding risk
Inter-practician variability of clinical care of venous thromboembolic according to patient body weight | up to 6 months after inclusion
  patient characteristics are : cancer, extreme body weight, severe renal impairment, elderly or pregnant patients, high bleeding risk
Inter-practician variability of clinical care of venous thromboembolic according to patient bleeding risk | up to 6 months after inclusion
  patient characteristics are : cancer, extreme body weight, severe renal impairment, elderly or pregnant patients, high bleeding risk

CONTACTS AND LOCATIONS:
Overall Officials: Simon Soudet, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No